CLINICAL TRIAL: NCT00005074
Title: A Phase II Study of Flavopiridol (HMR 1275; NSC 649890) in Patients With Untreated or Relapsed Mantle Cell Lymphoma
Brief Title: Flavopiridol in Treating Patients With Previously Untreated or Relapsed Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I127; CAN-NCIC-IND127 (Other: PDQ); NCI-100 (Other: NCI); CDR0000067679 (Other: PDQ)
Record Dates: First submitted 2000-04-06; First posted 2003-01-27 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Lymphoma
Keywords: stage I mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; stage II mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell | interventions — alvocidib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: alvocidib

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of flavopiridol in treating patients who have previously untreated or relapsed mantle cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the efficacy of flavopiridol in terms of response rate in patients with previously untreated or relapsed mantle cell lymphoma.
* Assess the toxicity of this regimen in this patient population.
* Determine the time to progression and, if responses are observed, response duration in these patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive flavopiridol IV over 1 hour daily for 3 days. Treatment continues every 3 weeks in the absence of unacceptable toxicity or disease progression. Patients with a complete response (CR) receive 2 additional courses after documented CR. Patients with a partial response receive 2 additional courses after documented maximal tumor shrinkage. Patients with stable disease receive a maximum of 4 courses.

Patients are followed at 4 weeks and then every 3 months until relapse or death.

PROJECTED ACCRUAL: A total of 14-30 patients will be accrued for this study within 18-24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed mantle cell lymphoma (at initial diagnosis) nonrefractory to prior therapy or with no prior therapy

  * No documented disease progression while receiving prior chemotherapy
* CD20 and CD5 positive
* Presence of clinically and/or radiologically documented disease
* At least 1 site of disease must be bidimensionally measurable

  * Bone lesions not considered bidimensionally measurable
  * Minimum indicator lesions must be:

    * Lymph nodes at least 1.5 cm x 1.5 cm by physical exam or spiral CT scan OR
    * Other nonnodal lesions at least 1 cm x 1 cm by MRI, CT scan, or physical exam
* No known CNS involvement by lymphoma

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute granulocyte count at least 1,500/mm3
* Platelet count at least 75,000/mm3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit or normal (ULN)
* AST no greater than 2.5 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No clinically significant cardiac symptomatology
* If history of cardiac disease, cardiac ejection fraction greater than 50%

Pulmonary:

* No clinically significant pulmonary symptomatology
* If history of symptomatic pulmonary disease:

  * FEV1, FVC, and TLC greater than 60% predicted
  * DLCO greater than 50% predicted

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Must be accessible for treatment and follow-up (i.e., no geographical limitations)
* No uncontrolled bacterial, fungal, or viral infection
* No other serious concurrent disease

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior radioactive monoclonal antibody therapy
* Prior rituximab allowed

Chemotherapy:

* See Disease Characteristics
* No more than 2 prior chemotherapy regimens allowed
* Same chemotherapy combination given for first line and second line therapy considered 2 regimens
* At least 6 weeks since prior chemotherapy
* No prior high-dose chemotherapy and stem cell transplantation
* No other concurrent cytotoxic chemotherapy

Endocrine therapy:

* No concurrent corticosteroids

Radiotherapy:

* No prior radiotherapy to greater than 25% of functioning bone marrow
* At least 4 weeks since prior radiotherapy (except low-dose, non-myelosuppressive radiotherapy) and recovered
* No concurrent radiotherapy to sole site of measurable disease

Surgery:

* At least 2 weeks since prior major surgery

Other:

* No other concurrent investigational anticancer agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2000-01-24 (Actual); Primary Completion 2002-02-20 (Actual); Study Completion 2008-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M. Connors, MD, Study Chair — British Columbia Cancer Agency
Locations (4):
- Canada (4):
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Humber River Regional Hospital, Weston, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kouroukis CT, Belch A, Crump M, Eisenhauer E, Gascoyne RD, Meyer R, Lohmann R, Lopez P, Powers J, Turner R, Connors JM; National Cancer Institute of Canada Clinical Trials Group. Flavopiridol in untreated or relapsed mantle-cell lymphoma: results of a phase II study of the National Cancer Institute of Canada Clinical Trials Group. J Clin Oncol. 2003 May 1;21(9):1740-5. doi: 10.1200/JCO.2003.09.057. PMID 12735303